CLINICAL TRIAL: NCT04561089
Title: Evaluation of the COVIDSeq Test in Saliva Specimens From Illumina Personnel
Brief Title: Evaluation of the COVIDSeq Test in Saliva Specimens From COVID-19 Asymptomatic Illumina Personnel
Status: Completed | Type: Observational
Sponsor: Illumina, Inc. (Industry)
Collaborators: Helix OpCo, LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: COVD-B07-001
Record Dates: First submitted 2020-09-21; First posted 2020-09-23 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva & nasal swab medium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 asymptomatic population: COVID-19 asymptomatic Illumina personnel
  Interventions: Diagnostic Test: COVIDSeq Test

INTERVENTIONS:
Diagnostic Test: COVIDSeq Test — The COVIDSeq is designed to test RNA extracted from NP swab specimens from patients symptomatic for COVID-19

SUMMARY:
"This is a prospective, multi-center specimen collection study. Subjects 18 years of age or older who do not have symptoms of COVID-19 will be enrolled. Two nasal swab samples and one saliva sample will be collected from each subject. The saliva sample will be tested with the COVIDSeq Test and one nasal swab will be tested with an EUA approved COVID test. The other nasal swab sample will be stored and a subset (approximately 250 specimens) will be tested with the COVIDSeq Test. Results of all testing will be provided to the sponsor for statistical analysis.

Positive results from COVIDSeq Test using saliva and/or the comparator EUA test will be provided to subjects so participants can be referred for further evaluation (outside the study). No medical treatment, guidance on treatment decisions, nor medical care will be provided. "

ELIGIBILITY:
Subject Inclusion Criteria:

An individual must meet the criteria below to be eligible.

* Individual is Illumina US personnel (eg, employee, contractor, consultant) and was invited to participate in the study.
* Individual is 18 years or older at the time of consent.
* Individual is feeling well and, at the time of consent or specimen collection, does not have any of the following symptoms of COVID-19: cough, shortness of breath or difficulty breathing, fatigue, fever or chills, muscle or body aches, headache, sore throat, new loss of taste or smell, congestion or runny nose, nausea or vomiting, or diarrhea. [1]
* Individual is willing to participate in study procedures and able to provide written informed consent in the English language.

Subject Exclusion Criteria:

An individual cannot meet the below criteria.

* Individual is confirmed to have COVID-19 and continues to require home isolation in accordance with current CDC guidelines at the time of consent or specimen collection.
* Individual is asymptomatic but suspected to have COVID-19 due to recent close contact (as currently defined by the CDC) with a person with COVID-19 and continues to require quarantine in accordance with current CDC guidelines at the time of consent or specimen collection. [4]
* Individual had symptoms of COVID-19 less than 10 days before time of consent or less than 10 days before time of any subsequent specimen collection visit."

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Illumina personnel
Sampling Method: Non-Probability Sample
Enrollment: 763 (Actual)
Dates: Start 2020-02-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Positive percent agreement (PPA) and negative percent agreement (NPA) between the COVIDSeq Test and a comparator EUA test for the detection of SARS-CoV-2 RNA | 1 month

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Illumina Laboratory Services, Foster City, California
  - Illumina Hayward, Hayward, California
  - Illumina Laboratory Services, San Diego, California